CLINICAL TRIAL: NCT06976346
Title: Pharmacokinetics and Relative Bioavailability Study of HRG2010 Capsule After Single Dose Administration
Brief Title: Relative Bioavailability Study of HRG2010 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HRG2010-101
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; benserazide, levodopa drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence A (Experimental): Period 1: HRG2010 dose 1 Period 2: HRG2010 dose 2 Period 3: Sinemet® Period 4: Madopar®
  Interventions: Drug: HRG2010 Capsule, Sinemet®, Madopar®
- Sequence B (Experimental): Period 1: HRG2010 dose 2 Period 2: Madopar® Period 3: HRG2010 dose 1 Period 4: Sinemet®
  Interventions: Drug: HRG2010 Capsule, Sinemet®, Madopar®
- Sequence C (Experimental): Period 1: Sinemet® Period 2: HRG2010 dose 1 Period 3: Madopar® Period 4: HRG2010 dose 2
  Interventions: Drug: HRG2010 Capsule, Sinemet®, Madopar®
- Sequence D (Experimental): Period 1: Madopar® Period 2: Sinemet® Period 3: HRG2010 dose 2 Period 4: HRG2010 dose 1
  Interventions: Drug: HRG2010 Capsule, Sinemet®, Madopar®

INTERVENTIONS:
Drug: HRG2010 Capsule, Sinemet®, Madopar® — In each period under fasting conditions, subjects received oral administration of either HRG2010 Capsule dose 1, HRG2010 Capsule dose 2, Sinemet®, or Madopar®.

SUMMARY:
This is a single-center, randomized, open-label, four-period, crossover study. Primary Objective：

1. To evaluate the pharmacokinetic characteristics of healthy subjects after a single oral dose of HRG2010 capsules at dose 1 and dose 2 under fasting conditions, and to compare these with the pharmacokinetic characteristics of Carbidopa/Levodopa Extended-Release Tablets (Sinemet®) and Benserazide/Levodopa Tablets (Madopar®).

   Secondary Objective
2. To assess safety following administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 18 and 45 years, inclusive.
2. At least 50.0 kg for male subjects, 45.0 kg for female subjects, with a Body Mass Index (BMI) between 19.0-26.0 kg/m2, inclusive (BMI = weight/height2).
3. Prior to screening, during the trial, and for 6 months after the trial, subjects (including male subjects) must not have plans to conceive and must voluntarily adopt effective contraceptive measures.
4. Subjects who could understand the nature, significance, potential benefits, inconvenience, and potential risks of the study, understand the procedures and methods, be willing to complete the trial strictly following the protocol, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Subjects with history of drug or food allergies.
2. Subjects with a history of diseases related to the circulatory, endocrine, nervous, digestive, respiratory, hematolymphatic, immune, mental, skin, bone, muscle, urogenital, mucosal, and metabolic systems, who are deemed by the investigator to be unsuitable for inclusion in this study.
3. Subjects with a history of glaucoma.
4. Use of any medication within 14 days prior to dosing.
5. Subjects who have taken any clinical investigational products or participated in the clinical research of medical devices within 3 months before the trial, or plan to participate in other clinical trials during the study.
6. Subjects who have donated blood or experienced blood loss greater than 300 mL, or have received a blood transfusion or used blood products within 3 months prior to screening, or plan to donate blood during the trial or within 1 month after the trial ends.
7. Subjects who had undergone major trauma surgery within 3 months before the screening, or planned a surgery during the study.
8. Subjects who take more than 5 cigarettes per day on average within 3 months prior to the study or do not agree to prohibit smoking during the study.
9. Drinking frequently within 6 months before the trial, meaning 14 units of alcohol per week（1 unit = 360 mL beer or 45 mL of 40% spirits, or 150 mL wine of 12% spirits), or disagree with the prohibition of alcohol during the study.
10. Clinical significance in clinical laboratory tests (chemistry, hematology, urinalysis, coagulation function).
11. Clinical significance in vital signs, physical examination, 12 lead-ECG.
12. Positive results in any one of Hepatitis B virus surface antigen, hepatitis C virus antibody, HIV antibody or syphilis serum reagin test.
13. Female who are pregnant or breastfeeding.
14. Breath test for alcohol > 0.0 mg /mL.
15. Subjects who were positive in drug abuse or had a history of drug abuse.
16. Difficulty in venous blood collection or unable to tolerate venipuncture or a history of fainting due to needle or blood phobia.
17. Subjects with swallowing difficulties, or those with special dietary requirements that prevent them from adhering to a unified diet.
18. Unable to complete the study due to personal reasons or other factors considered by the investigator as unsuitable to participate in the study (such as inability to understand the study requirements, poor compliance, etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum plasma concentration. Blood samples will be collected. | From 0 hour predose up to 12 hours postdose
AUC0-t: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected. | From 0 hour predose up to 12 hours postdose
AUC0-∞: Area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected. | From 0 hour predose up to 12 hours postdose
Tmax: Observed time to reach Cmax. Blood samples will be collected. | From 0 hour predose up to 12 hours postdose

SECONDARY OUTCOMES:
Incidence of treatment emergent AEs (TEAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 22)

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Province Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided